CLINICAL TRIAL: NCT02387021
Title: Prospective Comparison Between Continuous Femoral Nerve Block and the Association of Adductor Canal Block and Sciatic Nerve Block in Total Knee Arthroplasty.
Brief Title: Continuous Adductor Canal Block for Total Knee Arthroplasty Analgesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut Kassab d'Orthopédie (Other)
Responsible Party: Principal Investigator, Rais Karim, Dr, Institut Kassab d'Orthopédie
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P-2015002/AR
Record Dates: First submitted 2015-03-04; First posted 2015-03-12 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Neuromuscular Blockade; Pain Management
Keywords: analgesia; nerve block; Total knee replacement
MeSH Terms: conditions — Agnosia | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continous femoral nerve block (Active Comparator): Patients will receive ultrasound-guided (USG) continuous femoral nerve block with 20 ml ropivacaine 0.2% and USG Continuous adductor canal block with 20 ml of saline and USG infragluteal SNB with 20 ml of saline .
  Interventions: Procedure: Continuous femoral nerve block; Procedure: Continuous adductor canal block; Procedure: infragluteal Sciatic nerve block; Drug: Ropivacaine 0.2%; Drug: Saline
- Continuous adductor canal block (Experimental): Patients will receive ultrasound-guided continuous adductor canal block with 20 ml ropivacaine 0.2% and USG infragluteal SNB with 20 ml ropivacaine 0.2% and USG continuous FNB with 20 ml of saline .
  Interventions: Procedure: Continuous femoral nerve block; Procedure: Continuous adductor canal block; Procedure: infragluteal Sciatic nerve block; Drug: Ropivacaine 0.2%; Drug: Saline

INTERVENTIONS:
Procedure: Continuous femoral nerve block
Procedure: Continuous adductor canal block
Procedure: infragluteal Sciatic nerve block
Drug: Ropivacaine 0.2%
Drug: Saline

SUMMARY:
The purpose of the study is to determine whether the association of sciatic nerve block to continuous adductor canal block is effective in the treatment of total knee arthroplasty post operative pain .

ELIGIBILITY:
Inclusion Criteria:

* Elective unilateral TKA,
* Planned continuous spinal anesthesia ,
* Ability to follow study protocol,
* American Society of Anesthesiologists class 1 to 3.

Exclusion Criteria:

* Contraindication for neuraxial anesthetic,
* Chronic opioid use (defined as daily or almost daily use of opioids for >3 months),
* Hypersensitivity and/or allergies to any of the study medications,
* Intraoperative use of volatile anesthetics,
* Preexisting neuropathy on the operative limb,
* Contraindications to a femoral, adductor canal or Tibial nerve block.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Total Opioid-consumption | 8 hours postoperative
  Cumulative opioid consumption : converting oral, intravenous, and patient-controlled analgesia PCA opioid to morphine equivalent

SECONDARY OUTCOMES:
NRS pain score at rest | 0,1,2,4,6,8,12,24 and 48 hours postoperative
  NRS pain scores determined by patient interview, using the standard NRS of 0 to 10 scale at rest.
NRS pain score during movement | 0,1,2,4,6,8,12,24 and 48 hours postoperative
  NRS pain scores determined by patient interview, using the standard NRS of 0 to 10 scale, during physiotherapy.
NRS pain score after 10 meters of walk or maximum walked distance | 8, 24 and 48 hours postoperative
  NRS pain scores determined by patient interview, using the standard NRS of 0 to 10 scale after 10 meters walk (if enable after maximum walked distance).
Ability to walk | 8, 24 and 48 hours postoperative
  The ability of the patient to stand up and walk 3 meters.
TUG Test | 8, 24 and 48 hours postoperative
  The TUG test measures the time it takes a patient to stand up from a chair, walk a distance of 3 m, and return to the chair
The 10-m walk test | 8, 24 and 48 hours postoperative
  time it takes the patient to walk a distance of 10 m as quickly as possible
patient satisfaction | 8, 24 and 48 hours postoperative
  patient interviewed, using a scale of 0-10, 0 not satisfied and 10 being the most satisfied

REFERENCES:
- [Background] Kim DH, Lin Y, Goytizolo EA, Kahn RL, Maalouf DB, Manohar A, Patt ML, Goon AK, Lee YY, Ma Y, Yadeau JT. Adductor canal block versus femoral nerve block for total knee arthroplasty: a prospective, randomized, controlled trial. Anesthesiology. 2014 Mar;120(3):540-50. doi: 10.1097/ALN.0000000000000119. PMID 24401769